CLINICAL TRIAL: NCT00183079
Title: Brief Alcohol Intervention With Depressed Patients
Brief Title: Reducing Alcohol Use in Depressed Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAARAM13895; R01AA013895 (NIH); NIH 5 R01 AA13895
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2008-10

CONDITIONS: Depression; Alcohol Use
Keywords: Depression; Alcohol Use; Motivational Interviewing
MeSH Terms: conditions — Depression; Alcohol Drinking | interventions — Ethanol; Methods

ARMS (1):
- 1 (Active Comparator): Brief, motivationally-focused alcohol intervention
  Interventions: Behavioral: Motivationally-focused brief alcohol intervention

INTERVENTIONS:
Behavioral: Motivationally-focused brief alcohol intervention — Brief, motivationally-focused alcohol intervention

SUMMARY:
The purpose of this study is to determine whether a brief alcohol intervention reduces alcohol use and improves depression among depressed patients.

DETAILED DESCRIPTION:
Heavy alcohol consumption is common among patients seeking treatment for depression. Heavy drinking is associated with a variety of medical and psychosocial problems. Heavy drinking is particularly problematic among depressed patients, increasing the likelihood of poor depression treatment outcomes. While methods for reducing alcohol use in this population have been unexplored to date, brief interventions to reduce heavy alcohol use have been well-validated in numerous patient populations and offer the promise to reduce heavy drinking among depressed patients and to improve depression treatment outcomes.

We hypothesize that adding a brief alcohol intervention to standard psychiatric care, relative to standard psychiatric care alone, will reduce overall drinking volume and heavy drinking days among heavy-drinking depressed patients. Furthermore, we expect patients who receive the brief alcohol intervention to have better depression outcomes than patients receiving standard psychiatric care alone. We also expect that reduced alcohol consumption will mediate the effect of the brief alcohol intervention on depression outcomes. In addition, we will examine individual difference variables as predictors of change in alcohol use.

The proposed study is a randomized, two-group design with repeated measures over time, comparing a brief, motivationally-focused alcohol intervention plus standard psychiatric care to standard psychiatric care alone. For this study, we will recruit a sample of 240 psychiatry clinic outpatients meeting structured diagnostic criteria for major depressive disorder who drink heavily but are not alcohol dependent.

We expect that the results of this study will improve depression treatment outcomes for the significant subpopulation of depression patients who drink heavily and are likely to do poorly in depression treatment in the absence of a change in their drinking behavior. The intervention proposed in this study represents a novel approach to reducing heavy drinking among depressed patients that, if effective, can be readily integrated into depression treatment in a variety of treatment settings. In addition, this study will provide valuable information on the association between alcohol use and depression outcomes and on the mechanisms of change in alcohol use among heavy-drinking depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Meet criteria for current Major Depressive Disorder
* Have consumed more than 14 drinks per week or more than 5 drinks on one occasion in the past month for men or more than 7 drinks per week or more than 4 drinks on one occasion in the past month for females

Exclusion Criteria:

* Meet criteria for current alcohol dependence or current psychoactive substance dependence (excluding nicotine)
* Currently psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 6 months
Depressive symptoms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States